CLINICAL TRIAL: NCT00270582
Title: A Randomized Phase II Study of Weekly Docetaxel Plus Cisplatin Followed by Gemcitabine vs. Gemcitabine Plus Cisplatin Followed by Weekly Docetaxel in the Treatment of Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of Weekly Docetaxel Plus Cisplatin Followed by Gemcitabine vs. Gemcitabine Plus Cisplatin Followed by Weekly Docetaxel in the Treatment of Advanced Non-Small-Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-94015
Record Dates: First submitted 2005-12-26; First posted 2005-12-28 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2005-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: Taxotere, Cisplatin, Gemcitabine

SUMMARY:
Primary to evaluate the 1-year treatment failure rate of two sequential chemotherapy regimens:

1. weekly docetaxel plus cisplatin followed by gemcitabine and
2. gemcitabine plus cisplatin followed by weekly docetaxel. Study design:Prospective, multi-center, open-labelled, randomized phase II study.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in men and women worldwide. Shifting trends in the incidence of lung cancer closely follow the patterns of cigarette smoking, although other carcinogens have been implicated. Despite intensive over the past several decades, the 5-yr lung-cancer survival rate remains a dismal 8-14%.

Although lung cancer is not the most common cancer, as the leading cause of cancer-related deaths in men and women, it is the most deadly (American Cancer Society 2000). Lung cancer is also the leading cause of cancer deaths in Taiwan. According to the vital statistics of Department of Health in Taiwan, the incidence of lung cancer is rank of 5th. However, the rank of cancer fatality is the second and first in men and women, respectively. The mortality of lung cancer have significant increasing trend in men and women during the two-decade period. There are 6,555 persons die for lung cancer in 2001.

There is only 25% of cases resectable when diagnosed and only 15~18% of cases can be surgical removed. The postoperative recurrence rate and metastasis rate are also high for NSCLC. Chemotherapy is used primarily to palliate disease symptoms and prolong survival in patients with unresectable disease (stage IIIB and IV). However, overall survival benefit is modest.

Gemcitabine has shown good activity in NSCLC, both as a single agent and in combination with various other cytotoxic drugs (Eli Lilly and Company 1999). A number of phase I and II studies in NSCLC have shown good safety and efficacy of two-drug combinations of Gemcitabine with agents other than cisplatin, including carboplatin, paclitaxel, vinorelbine, and docetaxel (Eli Lilly and Company 1999).

Gemcitabine plus cisplatin (GC) is one of the most active regimens in the treatment fir stage IIIB/IV NSCLC patients. In phase II studies, 26-54% stage IIIB/IV NSCLC patients respond to GC treatment. Good median and 1-year survival have been consistently observed (Abratt et al, 1997; Crino et al, 1997; Einhorn, 1997; Shepherd et al, 1997) In randomized phase III studies, GC demonstrated the superior survival versus cisplatin alone (Sandler A et al. 2000), significantly higher response rate versus a three-drug combination of cisplatin, mitomycin C and ifosfamideb (Crino L et al. 1999).

Schiller JH et al. conducted a randomized study to determine whether any of three chemotherapy regimens was superior to cisplatin and paclitaxel in patients with advanced non-small-cell lung cancer (Schiller JH et al. 2000). Patients with advanced non-small-cell lung cancer were randomly assigned to a reference regimen of cisplatin and paclitaxel or to one of three experimental regimens: cisplatin and gemcitabine, cisplatin and docetaxel, or carboplatin and paclitaxel. However, none of four chemotherapy regimens offered a significant advantage over the others in the treatment of advanced non-small-cell lung cancer. GC provided longer time to progression than other three regimens.

Abratt et al (1997) used GC in stage IIIB/IV patients delivering cisplatin on day 15 resulted in goodresponse rate (52%), median survival (13 months) associated with low haematological toxicity and very few dose modifications of either gemicitabine or ciplatin. This schedule seems to be feasible for induction treatment.

Docetaxel plus cisplatin is one of options of front line treatment. TAX326- a phase III trial studied docetaxel + cisplatin or carboplatin vs vinorelbine/cisplatin (VC) as first-line therapy for advanced non-small cell lung cancer (NSCLC). The schedule of chemotherapy was 75 mg/m² of docetaxel followed by 75 mg/m² of cisplatin repeated every 3 weeks and Vinorelbine 25 mg/m2 IV day 1, 8, 15, 22 and Cisplatin 100 mg/m2 IV day 1 every 4 weeks. The overall response rate were 32% (docetaxel+cisplatin) and 25%(VC). Docetaxel plus cisplatin showed survival benefit compared to VC (1-year survival rate: 46% v.s. 41%).

Several phase II trials have investigated the efficacy and safety of Gemcitabine as a single agent, second-line therapy. Table below summarizes the results of the phase II trials.These trials concluded that gemcitabine has a modest activity as second-line chemotherapy for NSCLC. It has the advantage to be well tolerated and may thus be one drug to be proposed to the patients who have disease progression after a first-line chemotherapy and who ask for further treatment.

In the initial development of docetaxel and paclitaxel, these drugs routinely were administered once every 3 weeks. However, weekly administration of both these agents appears to offer several advantages in terms of toxicity. Both agents can be administered weekly with markedly decreased myelosuppression, while maintaining the same or increased dose intensity( Fennelly D et al 1997; Seidman AD et al 1998; Hainsworth JD et al 1998).

A Phase I trial demonstrated that docetaxel could be administered weekly at a maximum tolerated dose of 43 mg/m2/week, with fatigue and asthenia as the dose-limiting toxicities (Hainsworth JD et al 1998). At a weekly dose of 36 mg/m2, docetaxel was extremely well tolerated, with no significant myelosuppression and only occasional NCIC-CTG Grade 3 or 4 non-hematologic toxicities. The recommended dose was 36 mg/m2.

Four clinical studies of single-agent weekly docetaxel in patients with NSCLC have been reported. As second-line therapy for NSCLC, weekly docetaxel has been studied by 3 groups (Baylor-Charles 2000; Serke M et al 2001; Garcia-Lopez JL et al 2000 ), and Hainsworth JD and his colleagues studied weekly docetaxel as first-line treatment of NSCLC (Hainsworth JD et al 2000).

The 3 studies of weekly docetaxel as a single agent, second-line consistently demonstrated efficacy and similar toxicity profiles. Objective response rates ranged from 11% to 26.7%, and the percentage of patients who responded or maintained stable disease ranged from 37.5% to 66.7%. Docetaxel was generally well tolerated in each study.

Weekly docetaxel is being studied in combination with other commonly used NSCLC chemotherapeutic agents including carboplatin, navelbine, and gemcitabine. These combinations are being studied in both first- and second-line settings. Second line chemotherapy with docetaxel may affect survival (TAX 318, 1 year survival 37% vs. 11%). However, the optimal sequence of chemotherapy was rarely explored. Weekly docetaxel may offer better tolerability vs. 3-weekly schedule when combining docetaxel to cisplatin. Based upon these studied, we choose weekly docetaxel in combination with cisplatin as our regimen. We expected the regimen would be effective and well tolerated.

Based on the data above, this study proposed to compare the efficacy and safety of the two regimens (weekly docetaxel plus cisplatin followed by gemcitabine vs. gemcitabine plus cisplatin followed by weekly docetaxel) in metastatic of locally advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Written informed consent prior to beginning specific protocol procedures including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.

  2. Histologically or cytologically proven non-small cell lung carcinoma. 3. Stage IIIB or IV disease, no curative treatment available, candidate for chemotherapy.

  4. Age > 18 years and < 75 years. 5. Performance status WHO performance status 0,1. 6. Previous therapy:

  (a) Chemotherapy: None. (b) Previous radiation therapy : prior irradiation for NSCLC is permitted, however, the measurable or evaluable non-measurable disease must be completely outside the radiation portal.

  7. Unidimentional or bidimentional measurable disease. 8. Life expectancy > 12 weeks. 9. Laboratory requirements :
  1. Hematology: Neutrophils * 1.5 109/l, Platelets * 100 109/l, Hemoglobin > 10 g/dl.
  2. Hepatic function : Total bilirubin < 1.5 UNL, ASAT (SGOT) and ALAT (SGPT) < 2.5 UNL, Alkaline phosphatases < 5 UNL ; except in presence of only bone metastasis and in the absence of any liver disorders. Patients with ASAT and/or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study.
  3. Renal function : Creatinine < 1 UNL, and creatinine clearance should be > 60 ml/min.

     10.Complete initial lab studies within 2 weeks prior to first infusion, imaging studies within 4 weeks prior to first infusion.

     11.Patients must be accessible for treatment and follow-up.

     Exclusion Criteria:
* 1.Pregnant, or lactating patients; patients of childbearing potential must implement adequate contraceptive measures during study participation.

  2. Symptomatic central nervous system metastasis, patients with asymptomatic brain metastasis can be accepted if the tumor is irradiated and do not need steroid to control symptom.

  3. Pre-existing motor or sensory neurotoxicity of a severity > grade 1 by NCIC-CTG criteria.

  4. Other serious illness or medical condition :
  1. congestive heart failure or unstable angina pectoris. High risk uncontrolled arrhythmias.
  2. history of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
  3. active uncontrolled infection.
  4. contraindication for the use of corticosteroids. 5. Past or current history of neoplasm other than non small cell lung cancer, except for curatively treated non melanoma skin cancer, in situ carcinoma of the cervix within 5 years.

     6. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study entry.

     7. Concurrent treatment with any other anti-cancer therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2005-11

PRIMARY OUTCOMES:
To evaluate the 1-year treatment failure rate of two sequential chemotherapy regimens:
weekly docetaxel plus cisplatin followed by gemcitabine and
gemcitabine plus cisplatin followed by weekly docetaxel.

SECONDARY OUTCOMES:
To evaluate the median overall time to treatment failure (TTF).
To evaluate the overall progression free survival (PFS).
To evaluate the overall survival of each arm.
To evaluate the time to treatment failure for first regimen.
To evaluate the progression free survival for first regimen.
To evaluate the response rate for each regimen.
To evaluate the toxicity of each arm.
To evaluate the duration of response.

CONTACTS AND LOCATIONS:
Overall Officials: CHI HUANG HSIAO, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Chi-Huang Hsiao, Taipei, Ban-Ciao, Taiwan